CLINICAL TRIAL: NCT04968314
Title: ChiPP2: A Trauma-Informed Program for City School Parents
Acronym: ChiPP2
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Urban Health Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00232169
Record Dates: First submitted 2021-07-02; First posted 2021-07-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Parenting
Keywords: early childhood; adverse childhood events

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ChiPP Groups: Parents enroll in Chicago Parent Program groups offered at their child's school
  Interventions: Behavioral: Chicago Parent Program

INTERVENTIONS:
Behavioral: Chicago Parent Program — Chicago Parent Program (ChiPP) is a 12-session group-based parenting skills program

SUMMARY:
Purpose of this study is to assess the prevalence of adverse childhood experiences (ACEs) and positive childhood experiences (PCEs) among parents enrolled in the Chicago Parent Program (ChiPP) in their child's school and whether those experiences are associated with a) parents' participation in ChiPP and b) program benefits for parents and children.

DETAILED DESCRIPTION:
Purpose of this study is to assess the prevalence of adverse childhood experiences (ACEs) and positive childhood experiences (PCEs) among parents enrolled in the Chicago Parent Program (ChiPP) in their child's school and whether those experiences are associated with a) parents' participation in ChiPP and b) program benefits for parents and children. Parents who enroll in ChiPP groups in their child school are eligible to participate in this study. Data on ACEs, and PCEs are collected at baseline. Parent perceptions of their children's behavior problems and their engagement in early learning are collected at baseline and post-intervention data. Parent satisfaction with ChiPP and their sense of connection with other parents in their ChiPP group are measured at post-intervention only.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child enrolled in Chicago Parent Program group in Baltimore City Public Schools
* Parent age 18-99
* Child must be between 3-8 years old

Exclusion Criteria:

* Parent does not speak English or Spanish

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ChiPP is being offered in 11 Title 1 public schools in Baltimore and targets parents of young children (3-8 years old).
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Program participation | immediately after the intervention, approximately 4 months
  Number of Chicago Parent Program group sessions attended (range from 0-12 sessions)
Parent-reported child behavior frequency using the Eyberg Child Behavior Inventory | change from baseline to immediately after the intervention, approximately 4 months
  Parent-reported child behavior problems measured using the Eyberg Child Behavior Inventory. We will measure behavior problem frequency (scores range from 36-252). Higher scores indicate higher frequency.
Parent-reported child behavior problems using the Eyberg Child Behavior Inventory | change from baseline to immediately after the intervention, approximately 4 months
  Parent-reported child behavior problems measured using the Eyberg Child Behavior Inventory. We will measure whether the parent believes the behavior is a problem (scores range from 0-36). Higher scores indicate more child behavior problems.
Parent - Adverse childhood experiences | baseline
  number of adverse childhood experiences during parent's first 18 years of life assessed by parent report using the Philadelphia ACEs measure. Number of adverse childhood experiences assessed at baseline only. Includes two sub scales: the Conventional ACE sub scale (15 items measuring adversities in one's home) and the Expanded ACE sub scale (6 items measuring adversities in one's community). Scores can range from 0-21. Higher scores indicate more exposures to childhood adversity
Parent - Positive childhood experiences | baseline
  number of positive childhood experiences during parent's first 18 years of life assessed by parent-report at baseline using the Positive Childhood Experiences scale. Scores can range from 0-7 with higher scores indicating more exposures to positive childhood experiences.
Parent Satisfaction | immediately after the intervention, approximately 4 months
  Parent's satisfaction with the Chicago Parent Program intervention as assessed at post-intervention only and measured using the Chicago Parent Program Parent Satisfaction Form. Measure includes 19 items assessing the extent to which they and their child benefitted from the program (scored on a Likert-type scale), aspects of the program that were most and least beneficial, and the extent to which they would recommend the program to other parents. Each item is scored and interpreted separately.

SECONDARY OUTCOMES:
Social connectedness | immediately after the intervention, approximately 4 months
  parent-reported Likert-type measure of the extent to which parents developed a sense of connection and belonging with the other parents in the Chicago Parent Program intervention group. Measured using the 25-item Intervention Group Environment Scale and items are measured along a 5-point continuum of strongly disagree to strongly agree. Includes 3 sub scales measuring sense of belonging, quality of the group facilitation, and conflicts among members within the group. Scores can range from 0-5 with higher scores indicating greater social connectedness.
Parent engagement in early learning-Teacher Report | change from baseline to immediately after the intervention, approximately 4 months
  Measures teacher's perspective on the extent to which parents are engaged in their child's learning. Measured using a teacher-report measure (Teacher-Reported Parent Engagement in Child's Education) adapted from Fast Track measure of parent engagement. Teacher-Reported Parent Engagement in Child's Education includes 5 items assessed rated on a Likert-type scale; scores can range from 5-25 with higher scores indicating greater parent engagement from the perspective of the teacher. Measure completed by teachers.
Parent engagement in early learning-Parent Report | change from baseline to immediately after the intervention, approximately 4 months
  Measures the extent to which parents perceive they are engaged in their child's learning. Measured using the Parent Engagement in Early Childhood Education (PEECE) Survey. The PEECE Survey includes 25 items rated on a Likert-type scale. Scores can range from 25-100 with higher scores indicating greater engagement in their child's education.
Quality of parent participation in the intervention group | immediately after the intervention, approximately 4 months
  quality of each parent's participation in the Chicago Parent Program group sessions is assessed by group leaders using the Parent Engagement Rating Scale. This is a 7-item, 4-point Likert-type scale that assesses the extent to which the parent was actively engaged in the group sessions. Scores can range from 7-28 with higher scores indicating greater parent engagement and higher quality of participation in the group sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Gross, DNSc, Principal Investigator — Johns Hopkins University
Locations (1):
- Deborah Ann Gross, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Plesko CM, Yu Z, Tobin K, Richman R, Gross D. A mixed-methods study of parents' social connectedness in a group-based parenting program in low-income communities. Am J Orthopsychiatry. 2024;94(1):1-14. doi: 10.1037/ort0000695. Epub 2023 Oct 5. PMID 37796597